CLINICAL TRIAL: NCT03796000
Title: Characterization of Human Intestinal Macrophages in Metabolic Disease - iMAC (Pilot) Study
Brief Title: Characterization of Human Intestinal Macrophages in Metabolic Disease
Acronym: iMAC
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Claudia Cavelti, private lecturer, University Hospital, Basel, Switzerland
Other Study IDs: 2018-00712; 2018-00712 (Other: EKNZ)
Record Dates: First submitted 2018-12-21; First posted 2019-01-08 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- colonoscopy: obese and smoker: * 10 small tissue samples of the Colon transversum
  * 3 EDTA blood samples and 1 Serum blood sample
  * in some cases 1 single stool sample
  Interventions: Procedure: tissue samples, blood and stool sample
- colonoscopy: obese and non-smoker: * 10 small tissue samples of the Colon transversum
  * 3 EDTA blood samples and 1 Serum blood sample
  * in some cases 1 single stool sample
  Interventions: Procedure: tissue samples, blood and stool sample
- colonoscopy: lean and smoker: * 10 small tissue samples of the Colon transversum
  * 3 EDTA blood samples and 1 Serum blood sample
  * in some cases 1 single stool sample
  Interventions: Procedure: tissue samples, blood and stool sample
- colonoscopy: lean and non-smoker: * 10 small tissue samples of the Colon transversum
  * 3 EDTA blood samples and 1 Serum blood sample
  * in some cases 1 single stool sample
  Interventions: Procedure: tissue samples, blood and stool sample
- gastroscopy: obese and non-smoker undergoing bariatric surgery: * 6 small tissue samples of the gastric corpus and 6 of the Duodenum
  * 3 EDTA blood samples and 1 Serum blood sample
  * in some cases 1 single stool sample
  * 1cm long piece of the jejunum, which is usually disposed during bariatric surgery.
  Interventions: Procedure: tissue samples, blood and stool sample
- gastroscopy: lean and non-smoker: * 6 small tissue samples of the gastric corpus and 6 of the Duodenum
  * 3 EDTA blood samples and 1 Serum blood sample
  * in some cases 1 single stool sample
  Interventions: Procedure: tissue samples, blood and stool sample

INTERVENTIONS:
Procedure: tissue samples, blood and stool sample — Tissue samples from gastroscopy/colonoscopy.

SUMMARY:
This is a prospective, observational study aiming at improving the understanding of the pathophysiology of metabolic disease. As inflammation has been recognized as a key characteristic of metabolic disease but its starting point is still unknown, the investigators' aim is to characterize intestinal macrophages from human gut biopsies taken in diagnostic endoscopies of the gastrointestinal tract or in bariatric surgeries for clinical reasons.

DETAILED DESCRIPTION:
Metabolic disease including obesity and diabetes has reached epidemic proportions in the past years. Besides classical risk factors such as unhealthy diet and physical inactivity, smoking and air pollution have also emerged as unexpected risk factors for type 2 Diabetes.

Inflammation has been reported as key characteristic of metabolic disease and is predictive of future cardiovascular events. However, the starting point of chronic low-grade inflammation is not known.

As the gastrointestinal tract first comes into contact with dietary components, but potentially also air pollution/ smoke particles ingested upon mucociliary clearance from the lung, the gut could be the starting point of inflammation in metabolic disease.

The aim of this study is to characterize intestinal macrophages in obese versus lean subjects and smokers versus non-smokers to translate the principal investigator's preclinical findings to human disease and assess whether an inflammatory shift prevails in human intestinal macrophages in metabolic disease. Additionally, to assess whether intestinal macrophage subpopulations can be altered deliberately by nutritional intervention, the investigators will assess intestinal macrophages from subjects scheduled for bariatric surgery that will be on a calorie-restricted diet during the last 2 to 4 weeks prior to surgery.

The macrophages originate from human gut samples. As patients will undergo diagnostic endoscopy of the gastrointestinal tract or bariatric surgery for clinical reasons and the standard of care will not be changed by the study, there will be no additional interventions to patients by their participation in the study. Additionally, three EDTA and one serum blood tube for the analysis of inflammatory cells and markers in the blood will be taken as well as a single stool sample. The investigators' goal is to recruit in total 150 patients as it will be a pilot study in a first step.

ELIGIBILITY:
Inclusion Criteria:

Patient undergoing colonoscopy:

* Obese (BMI > 32 kg/m2 ) and smoker (≥ 1 pack cigarettes/d)
* Obese (BMI > 32 kg/m2 ) and non-smoker (control group)
* Lean (BMI < 27 kg/m2 ) and smoker (≥ 1 pack cigarettes/d)
* Lean (BMI < 27 kg/m2 ) and non-smoker (control group)

Patient undergoing gastroscopy:

* Obese (BMI > 35 kg/m2 ) and non-smoker planned for bariatric surgery
* Lean (BMI < 27 kg/m2 ) and non-smoker (control group)

Exclusion Criteria:

* Inability to provide informed consent, e.g. mental impairment or insufficient knowledge of project language
* Intake of corticosteroids
* Anti-inflammatory/ immunosuppressive drugs
* Clinical signs of current infection
* Known anemia (e.g. hemoglobin < 110 g/L for males, < 100 g/L for females)
* Known neutropenia (e.g. leukocyte count < 1.5 × 10^9/L or ANC < 0.5 × 10^9/L)
* Known immunodeficiency, e.g. HIV
* Known vasculitis, collagenosis
* Known inflammatory bowel disease
* Known adrenal insufficiency and/or substitution with glucocorticoids
* Known clinically significant kidney or liver disease (e.g. creatinine > 1.5 mg/dL, AST/ALT > 2 × ULN, alkaline phosphatase > 2 × ULN, or total bilirubin [tBili] > 1.5 × ULN)
* Risky daily alcohol consumption (> 24g/d for males, > 12g for females), known liver cirrhosis Child B or C
* Known uncontrolled congestive heart failure
* Known uncontrolled malignant disease
* Currently pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients planned for diagnostic endoscopy of the gastrointestinal tract or bariatric surgery at the University Hospital of Basel, the doctor's Office MagenDarm Basel or the Department of Visceral Surgery, Hospital Lindenhof of Bern will be screened for study participation, contacted and informed about the study if suitable to all inclusion and exclusion criterias.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-05-14 (Actual)

PRIMARY OUTCOMES:
Number of intestinal macrophages | 2 years
  Quantity (absolute and relative numbers) of intestinal macrophages in biopsies from the gastrointestinal tract in obese versus lean subjects and smokers versus non-smokers measured with flow cytometry.
Type and rate of subpopulations of intestinal macrophages | 2 years
  Quality (inflammatory versus non-inflammatory subpopulations) of intestinal macrophages in biopsies from the gastrointestinal tract in obese versus lean subjects and smokers versus non-smokers measured with flow cytometry.

SECONDARY OUTCOMES:
Number of other intestinal immune cells | 2 years
  In case the investigators do not find clear differences in frequency of intestinal macrophages, they will assess other intestinal immune cells (e.g. B-, T-lymphocytes), and enteroendocrine cells (e.g. L-cells) as a secondary endpoint in an explorative manner. Additionally, the investigators aim to correlate their findings from the biopsy samples with inflammation markers and immune cells in the blood, with microbiota and immune cells in the stool and with the eating habits of the patients.
Type and rate of subpopulations of other intestinal immune cells | 2 years
  In case the investigators do not find clear differences in subpopulations of intestinal macrophages, they will assess other intestinal immune cells (e.g. B-, T-lymphocytes), and enteroendocrine cells (e.g. L-cells) as a secondary endpoint in an explorative manner. Additionally, the investigators aim to correlate their findings from the biopsy samples with inflammation markers and immune cells in the blood, with microbiota and immune cells in the stool and with the eating habits of the patients.
Gene expression profile of intestinal macrophages | 2 years
  Gene expression of intestinal macrophages in biopsies from the colon in obese versus lean non-smokers by RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Cavelti-Weder, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT03796000/Prot_SAP_000.pdf